CLINICAL TRIAL: NCT06206291
Title: Cannabidiol in the Treatment of Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yasmin Hurd (Other)
Responsible Party: Sponsor-Investigator, Yasmin Hurd, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-21-00607; GCO# 21-0663 (Other Grant/Funding Number: National Institute On Drug Abuse/NIH/DHHS)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder
Keywords: CBD; Cannabidiol; Methadone; Buprenorphine; Opioid Use Disorder; OUD
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Methadone CBD (Active Comparator): CBD capsules (BSPG Laboratories) in two dosing periods for a total of 8 weeks.
  Interventions: Drug: Cannabidiol (CBD) 200mg; Drug: Cannabidiol (CBD) 400mg
- Methadone Placebo (Placebo Comparator): Matching placebo.in first dosing period and CBD 400mg in second dosing period
  Interventions: Drug: Placebo; Drug: Cannabidiol (CBD) 400mg
- Buprenorphine CBD (Active Comparator): CBD capsules (BSPG Laboratories) in two dosing periods for a total of 8 weeks.
  Interventions: Drug: Cannabidiol (CBD) 200mg; Drug: Cannabidiol (CBD) 400mg
- Buprenorphine Placebo (Placebo Comparator): Matching placebo.in first dosing period and CBD 400mg in second dosing period
  Interventions: Drug: Placebo; Drug: Cannabidiol (CBD) 400mg

INTERVENTIONS:
Drug: Placebo — Matching placebo twice daily for first 4 weeks
  Arms: Buprenorphine Placebo; Methadone Placebo
Drug: Cannabidiol (CBD) 200mg — First 4 weeks: CBD (200mg)/Placebo twice daily adjunct with opioid agonist treatment.
  Arms: Buprenorphine CBD; Methadone CBD
Drug: Cannabidiol (CBD) 400mg — Second 4 weeks: All cohorts receive CBD (400mg) twice daily adjunct with opioid agonist treatment.

SUMMARY:
The long-term goal of the project is to determine whether cannabidiol (CBD) can reduce craving and relapse in individuals with opioid use disorder (OUD). The first phase of our project was an open cross-over design study in healthy individuals to confirm the safety and pharmacokinetic (PK) effects of CBD. This next phase is to determine whether CBD can serve as a potential adjunct treatment to reduce craving and anxiety in individuals with OUD maintained on opioid agonist therapy.

DETAILED DESCRIPTION:
In this Phase 2 study, the research team will conduct a double-blind (placebo-controlled) randomized controlled trial to evaluate whether 200mg and/or 400mg CBD (BSPG Laboratories) given twice daily (morning and evening), as compared to placebo, reduces cue-induced craving and anxiety in individuals with opioid use disorder who are maintained on methadone or buprenorphine. In addition to in-lab physiological and behavioral assessments of cue-induced craving and anxiety, the research team will also employ ecological momentary assessment to obtain real-world measures of symptoms including craving, anxiety, and mood.

ELIGIBILITY:
INCLUSION CRITERIA:

An individual who meets all of the following criteria will be eligible for study participation:

* Individuals between 18 and 65 years old
* Ability to understand and give informed consent.
* Current opioid use disorder (OUD) or OUD in remission while on maintenance therapy with OAT, as determined by DSM-5 with the M.I.N.I. interview (Mini-International Neuropsychiatric Interview).
* Current opioid agonist maintenance treatment in an opioid treatment program with methadone or buprenorphine for at least 14 days prior to study participation. With the following more specific criteria for each of these two medications:

  * Current methadone maintenance treatment with a dose of ≥ 40mg/day, (maximum: 200mg/day), AND urinary toxicology positive for methadone and EDDP; OR
  * Current buprenorphine maintenance treatment with a dose of ≥ 8mg/day (maximum: 24mg/day), AND urinary toxicology positive for buprenorphine.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation:

* Participants who are non-English speaking.
* Psychiatric conditions under DSM-5 (examined with the MINI) that would make study participation unsafe or which would prevent adherence to study procedure; examples include: suicidal or homicidal ideation requiring immediate attention, inadequately-treated mental health disorder (e.g., active psychosis, uncontrolled bipolar disorder).
* Current diagnosis of a severe substance use disorder (except for opioid and nicotine/tobacco) in the past 3 months, based on the MINI interview, that would preclude safe participation in the study as determined by the study medical clinician.
* Alcohol intoxication when arriving at the study site (i.e., positive alcohol breathalyzer / alcohol salivary strips / urine alcohol).
* Signs of acute drug intoxication when arriving at the study site as determined by clinician assessment.
* Medical or psychiatric contraindications for CBD administration (e.g., history of hypersensitivity to cannabinoids); or any of the ingredients in the product (gelatin or sesame oil).
* Showing signs of acute opioid withdrawal symptoms (as determined by the result of the Clinical Opiate Withdrawal Scale (COWS). A Score of ≥ 5 or as interpreted by the investigator will be considered a positive result for withdrawal symptoms).
* Have a medical condition that would make study participation unsafe, which would make treatment compliance difficult, or would prevent adherence to study procedure. This includes, but is not limited to the following criteria:

  * History of impaired renal function or elevated liver enzymes at prescreening. The exclusionary lab values are: >4x the upper limit of normal (ULN) per laboratory criteria for AST or ALT, >1.5x ULN for bilirubin or <30mL/min/1.73m2 eGFR
  * QTc Frederica > 500ms
* Participating in another pharmacotherapeutic trial in the past 3 months.
* Participants who have used any medication, dietary supplements (and/or grapefruit juice), or combination of medications and supplements known to alter the metabolism of, or interact with CBD (buproprion, rifampin, barbiturates, phenothiazines, cimetidine, etc.) 14 days prior to and during the duration of the study
* For women: being pregnant (positive urine test for pregnancy) or breastfeeding.
* Not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e. condom, spermicide, diaphragm).
* Participants who have been court mandated to attend treatment centers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale for Craving (VASC) | Baseline and 4 weeks
  Cue-induced Visual Analog Scale for craving is used to measure subjective craving responses to a drug and neutral video cues evaluated in the clinic. Changes in craving from baseline (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Total scale ranges from 0-10, with higher scores indicating extreme cravings.
Change in Visual Analog Scale Anxiety (VASA) | Baseline and 4-weeks
  Cue-induced Visual Analog Scale Anxiety is used to measure subjective anxiety responses to a drug and neutral video cue evaluated in the clinic. Changes in anxiety from baseline (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Total scale from 0-10, with higher score indicating extreme anxiety.
Proportion of participants with positive urine toxicology | 4-weeks
  Proportion of participants with positive urine toxicology for illicit opioid use at 4 weeks.
Systematic Assessment for Treatment Emergent Events (SAFTEE) | weekly for 8 weeks
  Systematic Assessment for Treatment Emergent Events (SAFTEE) is used to measure safety and tolerability. SAFTEE is a side effect self-report assessment scale that consists of 56 potential side effects. Participants rate how bothersome each side effect is on a scale of "none" (0), "mild" (1), "moderate" (2), "severe" (3). Total score ranges 0 - 168, higher scores indicate a higher level of side effect burden.

SECONDARY OUTCOMES:
Change in Visual Analog Scale for craving (VASC) | baseline and 4-weeks
  Cue-induced Visual Analog Scale for craving is used to measure subjective craving responses to a drug and neutral video cues evaluated in the clinic. Changes in craving at 4 weeks compared to baseline (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Scale range: 0 (no craving) - 10 (extreme craving). Higher score indicates more extreme craving.
Change in Visual Analog Scale for craving (VASC) | 4-weeks and 8-weeks
  Cue-induced Visual Analog Scale for craving is used to measure subjective craving responses to a drug and neutral video cues evaluated in the clinic. Changes in craving at 8 weeks as compared to 4 weeks (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Scale range: 0 (no craving) - 10 (extreme craving). Higher score indicates more extreme craving.
Change in Visual Analog Scale Anxiety (VASA) | baseline and 4-weeks
  Cue-induced Visual Analog Scale Anxiety is used to measure subjective anxiety responses to a drug and neutral video cue evaluated in the clinic. Changes in anxiety at 4 weeks compared to baseline (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Scale: 0 (not at all anxious) - 10 (extremely anxious). Higher score indicates more extreme anxiety.
Change in Visual Analog Scale Anxiety (VASA) | 4-weeks and 8-weeks
  Cue-induced Visual Analog Scale Anxiety is used to measure subjective anxiety responses to a drug and neutral video cue evaluated in the clinic. Changes in anxiety at 8 weeks as compared to 4 weeks (pre-cue to post-cue and pre-neutral cue to post-neutral cue) will be measured and compared. Scale: 0 (not at all anxious) - 10 (extremely anxious). Higher score indicates more extreme anxiety.
Change in proportion of participants with positive urine toxicology | 4 weeks and 8 weeks
  Proportion of participants with positive urine toxicology for illicit opioid use at 8 weeks as compared to 4 weeks.
Change in Heroin Craving Questionnaire Short Form (HCQ-SF-14) | baseline and 4-weeks
  Heroin Craving Questionnaire Short Form (HCQ-SF-14): A 15 minute, 14 item self-administered to measure general heroin craving. Each item is rated on a 7-point Likert scale (1= strongly disagree, 7= strongly agree). Full scale ranges from 14-98, with higher scores indicating more severe heroin craving.
Change in Heroin Craving Questionnaire Short Form (HCQ-SF-14) | 4-weeks and 8-weeks
  Heroin Craving Questionnaire Short Form (HCQ-SF-14): A 15 minute, 14 item self-administered to measure general heroin craving. Each item is rated on a 7-point Likert scale (1= strongly disagree, 7= strongly agree). Full scale ranges from 14-98, with higher scores indicating more severe heroin craving.
Change in Generalized Anxiety Disorder Scale (GAD-7) | baseline and 4-weeks
  The General Anxiety Disorder 7-item questionnaire (GAD-7) assesses seven problem items potentially experienced over the past two weeks from "0" (not at all) to "3" (nearly every day). Individuals rank their levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more anxiety symptoms.
Change in Generalized Anxiety Disorder Scale (GAD-7) | 4-weeks and 8-weeks
  The General Anxiety Disorder 7-item questionnaire (GAD-7) assesses seven problem items potentially experienced over the past two weeks from "0" (not at all) to "3" (nearly every day). Individuals rank their levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more anxiety symptoms.
Duration of participant first illicit opioid abstinence | any time during study, 8 weeks
Change in Patient Health Questionnaire (PHQ-9) | baseline and 4-weeks
  The Questionnaire Type 9 for Depression (PHQ-9) measures depression severity with the nine DSM-IV criteria scored as "0" (not at all) to "3" (nearly every day). Full scale ranges from 0-27, with higher score indicating more severe symptoms.
Change in Patient Health Questionnaire (PHQ-9) | 4-weeks and 8-weeks
  The Questionnaire Type 9 for Depression (PHQ-9) measures depression severity with the nine DSM-IV criteria scored as "0" (not at all) to "3" (nearly every day). Full scale ranges from 0-27, with higher score indicating more severe symptoms.
Positive and Negative Affect Schedule (PANAS-SF) | baseline and 4-weeks
  A 20 item self-administered questionnaire evaluating current positive and negative affect. Each item is rated on a 5-point scale (0= Very slightly or not at all, 5= Extremely). Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.
Positive and Negative Affect Schedule (PANAS-SF) | 4-weeks and 8-weeks
  A 20 item self-administered questionnaire evaluating current positive and negative affect. Each item is rated on a 5-point scale (0= Very slightly or not at all, 5= Extremely). Scores range from 10 - 50 for both sets of items. For the total positive score, a higher score indicates more of a positive affect. For the total negative score, a lower score indicates less of a negative affect.
Change in Heart rate | baseline and 8-weeks
  Heart rate (beats/min) will be monitored throughout the time course of the study and changes from baseline will be studied.
Change in Blood pressure | baseline and 8-weeks
  Blood pressure (in mmHg) will be monitored throughout the time course of the study and changes from baseline will be studied. Both diastolic and systolic pressures will be assessed.
Change in Body Temperature | baseline and 8-weeks
  Body temperature (in degrees Fahrenheit) will be monitored throughout the time course of the study and changes from baseline will be studied.
Change in Oxygen level | baseline and 8-weeks
  Oxygen level will be measured by pulse oximetry when vitals are collected for each participant throughout the study.
Change in Cue-induced salivary cortisol levels | baseline and 4-weeks
  Study participant will chew on a cotton swab providing a saliva sample from which free cortisol levels will be measured as an indicator of stress response in association with video cues. Thus, the stress of craving will be monitored and measured to observe any changes from baseline.
Change in Cue-induced salivary cortisol levels | 4-weeks and 8-weeks
  Study participant will chew on a cotton swab providing a saliva sample from which free cortisol levels will be measured as an indicator of stress response in association with video cues. Thus, the stress of craving will be monitored and measured to observe any changes from 4-weeks.
Sleep duration | up to 8-weeks
  Average sleep duration measured across 8 weeks.
Change in Insomnia Severity Index (ISI) | baseline and 8-weeks
  A 5-10 minute, 7 question self-administered screening tool for insomnia. Each item rates the nature and symptoms of potential sleep problems using a 5-point Likert-type scale. Minimum score of 0 and maximum score of 28, with the highest score indicating prevalence and severity of insomnia.
Change in The Digit Span Test subtest of the Wechsler Adult Intelligence Scale 4th edition | baseline and 8-weeks
  A 10-15 minute 30-item assessment that includes Digit Span Forward (DSF) and Digit Span Backward (DSB). DSF measures short-term memory, not working memory. DSB measures auditory working memory. Full scale from a minimum score of 0 and maximum score of 30, with the highest score indicating the total number of points achieved for correct responses.
Change in The Symptom Check List 90 (SCL-90) | baseline and 8-weeks
  The Symptom Check List 90 (SCL-90): A 12-15 minute, 90 item self-administered psychometric instrument yielding nine scores of primary symptom dimensions (5-point rating scale; 1= Not at all, 5= Extremely), along with three scores based on global distress measures. Full scale ranges from a minimum score of 90 and maximum score of 450, with higher scores indicating more severe psychological distress.
Change in Substance use other than opioids in urine | baseline and 4-weeks
  Substance use other than opioids measured in urine.
Change in Substance use other than opioids in urine | 4-weeks and 8 weeks
  Substance use other than opioids measured in urine.
Change in Substance use other than opioids in blood | baseline and 4-weeks
  Substance use other than opioids measured in blood.
Change in Substance use other than opioids in blood | 4-weeks and 8 weeks
  Substance use other than opioids measured in blood.
Change in Concentration of methadone or buprenorphine metabolites in urine | baseline and 4-weeks
  Concentration of methadone or buprenorphine metabolites measured in urine.
Change in Concentration of methadone or buprenorphine metabolites in urine | 4-weeks and 8-weeks
  Concentration of methadone or buprenorphine metabolites measured in urine.
Change in Concentration of methadone or buprenorphine metabolites in blood | baseline and 4-weeks
  Concentration of methadone or buprenorphine metabolites measured in blood.
Change in Concentration of methadone or buprenorphine metabolites in blood | 4-weeks and 8-weeks
  Concentration of methadone or buprenorphine metabolites measured in blood.
Number of participants remaining in treatment | up to 8 weeks
  Retention in treatment
Change in Change in dosage of opioid agonist treatment | baseline and 8 weeks
Number of positive urine toxicology | 4 weeks
  The number of positive urine toxicology to measure adherence
Number of positive blood toxicology | 4 weeks
  The number of positive blood toxicology to measure adherence

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available, if the plan changes, the research team will share the plan details.

DOCUMENTS (1):
  • Informed Consent Form (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT06206291/ICF_000.pdf